CLINICAL TRIAL: NCT05184517
Title: A Feasibility, Double Blind, Randomized, Crossover Study to Evaluate the Tolerability of Oph1 0.5% Cyclosporine Ophthalmic Formulation Compared to Restasis in Healthy Volunteers
Brief Title: A Feasibility Study to Evaluate the Tolerability of Oph1 Compared to Restasis in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: OphRx Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CD-001
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded, participant and Outcome Assessors are blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (Experimental): Oph1 0.5% CsA ophthalmic formulation followed by Restasis 0.05% CsA ophthalmic formulation
  Interventions: Drug: Oph1; Drug: Restasis
- Arm II (Experimental): Restasis 0.05% CsA ophthalmic formulation followed by Oph1 0.5% CsA ophthalmic formulation
  Interventions: Drug: Oph1; Drug: Restasis

INTERVENTIONS:
Drug: Oph1 — 0.5% CsA ophthalmic formulation, twice daily for 4 days and once on the fifth day, one eye (right).
Drug: Restasis — 0.05% CsA ophthalmic formulation twice daily for 4 days and once on the fifth day, one eye (right).

SUMMARY:
20 healthy participants will be evaluated for tolerability and safety of a new eye drop formulation for treatment of Dry Eye Syndromes, Oph1 0.5% Cyclosporine A (CsA) compared with Restasis 0.05% CsA ophthalmic formulation.

DETAILED DESCRIPTION:
20 healthy participants will be enrolled to the study and randomized into two groups of 10 participants each. In one group participants will be treated with Oph1 0.5% CsA ophthalmic formulation and in the other group with Restasis 0.05% CsA ophthalmic formulation. Both groups will be treated with the eye drops in the right eye only, twice a day (6-9 hours apart), for four days and once on the fifth day (total of 9 eye drops treatment for each), both groups will have 2 days of washout, and will be crossed to identical course of treatment with the other ophthalmic formulation. All eye drops treatments will be done on the medical site by one of the study staff unblinded to the treatment. The Investigator assessing the ocular signs and the participants will be blinded to study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 20-50 years, inclusive.
2. Systemically and ophthalmologically healthy subjects evaluated during the clinical history.
3. Best-corrected visual acuity (BCVA) 20/40 or better in both eyes.
4. Negative Fluorescein staining in Fluorescein Corneal staining (FCS) in both eyes.
5. Up to 0.5 Conjunctival redness in Conjunctival redness without slit lamp, in standardized lighting conditions, in both eyes.
6. IOP (< 22mmHg), in both eyes.
7. No pathology findings in Slit-lamp biomicroscopy in both eyes.
8. Ability to comply with the requirements of the study and complete the questionnaire and a full sequence of protocol-related evaluations.
9. Ability to understand and provide written informed consent.
10. In the judgement of the investigator, the participant can safely perform study activity.

Exclusion Criteria:

1. Have chronic systemic disease of any form known.
2. In the case of women: be pregnant, breastfeeding or planning to become pregnant within the study period or women without a history of hysterectomy, oophorectomy, who do not ensure a hormonal contraceptive method or intrauterine device during the study period.
3. Be a user of topical ophthalmic products of any kind.
4. Being a chronic drug user.
5. Be a user of contact lenses.
6. Have a history of any type of eye surgery.
7. Participating in clinical research studies 90 days prior to inclusion in the present study.
8. In the judgement of the investigator, any condition that could interfere with the intent of the study or would make participation not in the best interest of the participant.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Drop Discomfort VAS score | up to Fifth day per treatment (last dose for each treatment)
  Eye Discomfort VAS scale from 0-100

SECONDARY OUTCOMES:
Drop Comfort VAS score | 1-minute post-Dose. Fifth day per treatment (last dose for each treatment)
  Eye Discomfort VAS scale from 0-100
Drop Discomfort Detailed VAS score. Calculated mean of all scores per treatment for each of the VAS scale. | 1 minutes post-Dose instillation, Day 1-5, Day 8-12, AM
  Eye Discomfort, Itching, Burning, Foreign body feel VAS scales from 0-100
Drop Discomfort Detailed VAS score. Calculated mean of all scores per treatment for each of the VAS scale. | 5 minutes post-Dose instillation, Day 1-5, Day 8-12, AM
  Eye Discomfort, Itching, Burning, Foreign body feel VAS scales from 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel